CLINICAL TRIAL: NCT05330299
Title: Acceptability of Identifying and Managing Psychological Distress in Inflammatory Bowel Disease: the COMPASS-IBD Study
Acronym: COMPASS-IBD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); Crohn's and Colitis UK (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 312818
Record Dates: First submitted 2022-03-18; First posted 2022-04-15 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-03

CONDITIONS: IBD; Psychological Distress; Treatment of Illness-related Distress in IBD

STUDY DESIGN:
Intervention Model Description: Participants will receive COMPASS as part of standard care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COMPASS (single arm) (Experimental): Participants will be treated with an online CBT program that is specifically tailored to illness-related distress in the context of IBD.
  Interventions: Behavioral: COMPASS

INTERVENTIONS:
Behavioral: COMPASS — Participants will be treated with an online CBT program that is specifically tailored to illness-related distress in the context of long-term conditions. It consists of 11 online modules and is therapist-supported.

SUMMARY:
This study is a single-centre, interventional implementation and feasibility study.

Patients in the IBD service will be able to access COMPASS, an online cognitive-behavioural therapy (CBT) programme, as part of standard care at Guy's and St Thomas's NHS Foundation Trust.

COMPASS is an online program. It will consist of 11 online modules which target challenges associated with living with IBD (and other long-term conditions) and includes, amongst other things, psycho-education, patient examples, interactive tasks and goal setting. Participants are linked to a therapist; 'guide', who will provide 5-6 x 30 minute support sessions delivered fortnightly in the format preferred by the client (phone and/or in-site message).

ELIGIBILITY:
PATIENT PARTICIPANTS

Inclusion Criteria:

1. Aged 18 or over
2. Have an IBD diagnosis
3. Have English proficiency
4. Have access to a computer
5. Have mild to moderate symptoms of depression and/or anxiety (PHQ-9 score 5-19 and/or GAD-7 score 5-14, or PHQ-ADS score 10-29) or severe depression and/or anxiety (PHQ-9 score≥20 and/or GAD-7 score ≥15, or PHQ-ADS score ≥30 but no acute suicidal risk) and awaiting treatment from clinical psychologist as specified above.
6. Have evidence of illness-related distress

Exclusion Criteria:

1. Evidence of substance dependency, cognitive impairment, severe mental health conditions
2. Evidence of acute suicidal risk PHQ-9 item-9 >1 and recent serious suicidal intent and/or planning
3. Are receiving current psychological treatment or are on a wait-list to receive treatment within the study period (next 6 months)
4. Have depression and/or anxiety unrelated to IBD (e.g. where disease long-standing/well-controlled unrelated to current presentation of distress)

HEALTHCARE PROFESSIONAL PARTICIPANTS

1. Work in the Gastroenterology IBD service at Guy's and St Thomas' Hospitals NHS Trust (GSTT).
2. Have experience of either: i) Utilising the routine mental health screening tools ii) Assessing and triaging patients onto the COMPASS programme and/or iii) Providing therapist support to the users of COMPASS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
The number and demographics of people who agree to and complete routine screening for psychological distress (including e-IMPARTS). | 18 months
  Assessing clinical reach of routine screening and the COMPASS intervention
The demographic characteristics of patients with IBD who report clinical levels of anxiety (according to IMPARTS pre-determined cut-offs) during routine mental health screening. | 18 months
  Assessing clinical reach of routine screening and the COMPASS intervention. Anxiety is measured with the Generalised Anxiety Disorder Scale (GAD-7). Min score = 0, Max score = 21, with higher scores indicating greater anxiety.
The proportion of patients with IBD who report clinical levels of anxiety (according to IMPARTS pre-determined cut-offs) during routine mental health screening. | 18 months
  Assessing clinical reach of routine screening and the COMPASS intervention. Anxiety is measured with the Generalised Anxiety Disorder Scale (GAD-7). Min score = 0, Max score = 21, with higher scores indicating greater anxiety.
The demographic characteristics of patients with IBD who report clinical levels of depression (according to IMPARTS pre-determined cut-offs) during routine mental health screening. | 18 months
  Assessing clinical reach of routine screening and the COMPASS intervention. Depression is measured with the Patient Health Questionnaire (PHQ-9). Min score = 0, Max score = 27, with higher scores indicating greater depression.
The proportion of patients with IBD who report clinical levels of depression (according to IMPARTS pre-determined cut-offs) during routine mental health screening. | 18 months
  Assessing clinical reach of routine screening and the COMPASS intervention. Depression is measured with the Patient Health Questionnaire (PHQ-9). Min score = 0, Max score = 27, with higher scores indicating greater depression.
The demographics of IBD patients who report clinical levels of psychological distress in the mild to moderate (PHQ-ADS distress score 10-29) and severe (PHQ-ADS distress score ≥30, but no acute suicidal risk) range at screening | 18 months
  Assessing clinical reach of routine screening and the COMPASS intervention. Psychological Distress is measured with the Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS). The PHQ-ADS is a composite measure of Generalised Anxiety Disorder questionnaire (GAD-7) and Patient Health Questionnaire (PHQ-9). Min score = 0, Max score = 48, with higher scores indicating higher levels of distress.
The proportion of IBD patients who report clinical levels of psychological distress in the mild to moderate (PHQ-ADS distress score 10-29) and severe (PHQ-ADS distress score ≥30, but no acute suicidal risk) range at screening | 18 months
  Assessing clinical reach of routine screening and the COMPASS intervention. Psychological Distress is measured with the Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS). The PHQ-ADS is a composite measure of Generalised Anxiety Disorder questionnaire (GAD-7) and Patient Health Questionnaire (PHQ-9). Min score = 0, Max score = 48, with higher scores indicating higher levels of distress.
Descriptive statistics of functioning in IBD patients, using the Work and Social Adjustment Scale questionnaire measured as part of standard care / routine screening. | 18 months
  Assessing clinical reach of routine screening and the COMPASS intervention. The Work and Social Adjustment Scale (WSAS) measures impaired functioning. Min score = 0, max score = 40, with higher scores indicating greater impaired functioning.
Descriptive statistics of control of IBD in IBD patients, using the IBD control questionnaire measured as part of standard care / routine screening. | 18 months
  Assessing clinical reach of routine screening and the COMPASS intervention. The IBD control measures the extent to which patients have control over their IBD. Min score = 0, max score = 16, with higher scores indicating poorer control.
The proportion of IBD patients who show evidence of acute suicidal risk at screening | 18 months
  Assessing clinical reach of routine screening and the COMPASS intervention
The demographic and clinical characteristics, and proportion of IBD patients who meet inclusion criteria and are willing and able to engage in the COMPASS treatment. | 18 months
  Assessing clinical reach of the COMPASS intervention
The reasons for study ineligibility (descriptively). | 18 months
  Assessing clinical reach of the COMPASS intervention. Descriptive data, specifically frequencies documenting the number of individuals who are willing to use COMPASS, reasons documented for ineligibility/non-uptake and the sociodemographic and clinical profile of eligible vs non-eligible of COMPASS.
COMPASS engagement | 18 months
  Assessing clinical reach of the COMPASS intervention. Descriptive data regarding demographic and clinical characteristics of non-engagers, less-adherent users and adherent-users of COMPASS.
Change in Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS) from pre- to post-treatment in IBD patients who receive COMPASS. | At baseline, 12 weeks (post-therapy), 6 months (follow-up)
  The PHQ-ADS will be used to establish the efficacy of treatment pathways for IBD patients. It is a composite measure of the Generalised Anxiety Disorder questionnaire (GAD-7) and the Patient Health Questionnaire (PHQ-9). Min score = 0, Max score = 48, with higher scores indicating higher levels of distress.
Change in Patient Health Questionnaire - (PHQ-9) | At baseline, 12 weeks (post-therapy), 6 months (follow-up)
  Depression. Min score = 0, Max score = 27, with higher scores indicating greater depression.
Change in Generalised Anxiety Disorder scale (GAD-7) | At baseline, 12 weeks (post-therapy), 6 months (follow-up)
  Anxiety. Min score = 0, Max score = 21, with higher scores indicating greater anxiety
Change in EQ-5D-3L | At baseline, 12 weeks (post-therapy), 6 months (follow-up)
  Quality of life. Min score = 5, Max score = 15 , with higher scores more problems in the scale dimensions.
Change in the The UK Inflammatory Bowel Disease Questionnaire (IBDQ-UK) | At baseline, 12 weeks (post-therapy), 6 months (follow-up)
  IBD-related Quality of Life. Min score = 0, Max score = 96. Higher values indicate better quality of life.
Change in the Patient Global Impression Scales of Severity (PGI-S) | At baseline, 12 weeks (post-therapy), 6 months (follow-up)
  Perceived symptom severity. 1 item. Min = 0, Max = 3, with higher scores indicating greater perceived symptom severity.
Change in the Brief Illness Perception Questionnaire (BIPQ) | At baseline, 12 weeks (post-therapy), 6 months (follow-up)
  Illness perceptions. Questionnaire adapted to use first 8 items: illness consequences and timeline, the controllability of the illness personally and through treatment, illness identity, concerns, coherence, and the emotional-impact of the illness. Each item on the BIPQ is assessed as a separate construct (for each construct, min = 0, max = 10). Higher scores relate to stronger/greater illness perceptions.
Change in the short Cognitive Behavioural Responses Questionnaire (CBRQ-short) | At baseline, 12 weeks (post-therapy), 6 months (follow-up)
  Views and behaviours regarding symptoms. Only 3 subscales will be used: embarrassment avoidance (3 items), symptom focusing (3 items) and all-or-nothing behaviour (3 items) subscales. Min = 0, Max = 36. Higher scores indicate poorer cognitive and behavioural responses.
Change in the Chronic Disease Self-efficacy Scale | At baseline, 12 weeks (post-therapy), 6 months (follow-up)
  Disease self-efficacy. 9 sub-scales will be used: exercise regularly, get information about disease, obtain help from community, communicate with physician, manage disease in general, do chores, social/recreational activity, manage symptoms, control/manage depression. Min scores = 0, Max scores = 320. Higher scores indicate higher self-efficacy.
Change in the Acceptance of Chronic Health Conditions Scale | At baseline, 12 weeks (post-therapy), 6 months (follow-up)
  Acceptance of illness. Min score = 0, Max = 40. Greater scores indicate higher levels of acceptance.
Change in Health Service Use Questionnaire | At baseline, 12 weeks (post-therapy), 6 months (follow-up)
  4 service use items (GP, psychologist, emergency care, secondary care service) from the client service receipt inventory (CSRI) will be used. Frequency and duration of particular services will be recorded, from which a total time will be calculated. There is no maximum value. Higher scores indicate more health service time used.
Change in Body Mass Index (BMI) | At baseline, 12 weeks (post-therapy), 6 months (follow-up)
  Weight (in kg) and Height (in m) will be combined to calculate BMI (weight in kg / (height in m)^2
Change in smoking status | At baseline, 12 weeks (post-therapy), 6 months (follow-up)
  Current smoking status, including amount of cigarettes consumed per day.
Change in alcohol consumption | At baseline, 12 weeks (post-therapy), 6 months (follow-up)
  Number of units drunk in the past week.
Change in the International Physical Activity Questionnaire | At baseline, 12 weeks (post-therapy), 6 months (follow-up)
  Physical activity. There are three subscales (vigorous activity, moderate activity and lower-level activity). Scores will be in minutes. Higher scores will indicate more physical activity performed.
Change in IBD activity | At baseline, 12 weeks (post-therapy), 6 months (follow-up)
  For Crohn's Disease patients: The Patient-Reported Outcomes for the Assessment of Crohn's Disease Activity (PRO-CD). The scale contains two sub-scales: 1) bowel signs and symptoms, 2) functional symptoms. Each scale is scored separately. There is no total score for the PRO-CD. The first sub-scale starts at 0 and has no maximum value, with greater scores indicating greater bowel signs/symptoms. The second subscale ranges from 0-21, with higher scores indicating greater functional symptoms.
  For Ulcerative Colitis / unclassified patients: The Patient-Reported Outcomes for Assessment of Ulcerative Colitis (PRO-UC). The scale has 9-items and includes two scales: 1) Bowel signs/symptoms and 2) functional symptoms. The first sub-scale starts at 0 and has no maximum value, with greater scores indicating greater bowel signs/symptoms. The second subscale ranges from 0-21, with higher scores indicating greater functional symptoms.
Change in IBD medication | At baseline, 12 weeks (post-therapy), 6 months (follow-up)
  Current medication and dose.
Change in IBD flares | At baseline, 12 weeks (post-therapy), 6 months (follow-up)
  Frequency and severity (4-point scale) of IBD flares
The Patient Global Impression Scales of Severity (PGI-S) | Baseline, 12 weeks (post-therapy), 6 months (follow-up)
  Perceived symptom severity. 1 item. Min = 0, Max = 3, with higher scores indicating greater perceived symptom severity.
The Patient Global Impression Scales of Improvement (PGI-I) | 12 weeks (post-therapy), 6 months (follow-up)
  Perceived symptom improvement. 1 item. Min = 0, Max = 6, with higher scores indicating greater perceived symptom deterioration.
The demographic characteristics of IBD patients who receive COMPASS while on the IBD psychology wait-list, but are removed from the wait-list at the end of COMPASS. | 18 months
  Descriptive data pertaining to demographics and frequencies. These data will be used to establish the efficacy of treatment pathways for IBD patients.
The clinical characteristics of IBD patients who receive COMPASS while on the IBD psychology wait-list, but are removed from the wait-list at the end of COMPASS. | 18 months
  These data will be used to establish the efficacy of treatment pathways for IBD patients.
The adoption of routine screening and the COMPASS programme. | For patients -12-weeks (post-therapy); For HCPs (over 18 months)
  Qualitative exploration the perspectives of healthcare professionals (HCPs) and patients
Scores in the NoMAD (tool for measuring implementation processes) as rated by healthcare professionals (HCPs) | 18 months
  23-item instrument for measuring implementation processes, organised by the Normalisation Process Theory framework.
The number of patients who require digital support to use COMPASS. | 18 months
  Exploration of the adoption of COMPASS
The change in numbers on and duration of the wait-list to see clinical psychologist from pre- to post-COMPASS | 18 months
  Exploration of the adoption of COMPASS
Patient adherence to online sessions | 12-weeks (post therapy)
  Adherence defined as 5 online sessions completed. Will be used to assess the implementation of COMPASS into the service.
Number and duration of therapist calls attended. | 12-weeks (post therapy)
  Adherence defined as 3 calls/messages attended.
Drop out rate of COMPASS | 18 months
  The number and proportion of patients that drop out of COMPASS will be recorded to assess the implementation of COMPASS into the service.

CONTACTS AND LOCATIONS:
Overall Officials: Rona Moss-Morris, PhD, Principal Investigator — King's College London
Locations (1):
- Health Psychology Section, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available on request from the corresponding author. The data will not be available publicly due to privacy or ethical restrictions.
Supporting Information: Study Protocol, ICF
Access Criteria: The data will only be available on request.

REFERENCES:
- [Derived] Jones ASK, Harding S, Seaton N, Hudson JL, Duff A, Wroe A, Singh H, Norton S, Picariello F, Moss-Morris R. A real-world longitudinal study implementing digital screening and treatment for distress in inflammatory bowel disease (IBD): The COMPASS-IBD study protocol. Contemp Clin Trials. 2024 Oct;145:107658. doi: 10.1016/j.cct.2024.107658. Epub 2024 Aug 8. PMID 39121990